CLINICAL TRIAL: NCT03916315
Title: Effectiveness of the Transdiagnostic Treatment in the Population of Tijuana and Juarez With Anxiety and Electrophysiological Correlation Measurements. A Randomized Clinical Trial
Brief Title: Transdiagnostic Treatment for Anxiety Disorders in Two Cities of México
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Baja California (Other)
Collaborators: Universidad Autonoma de Ciudad Juarez (Other)
Responsible Party: Principal Investigator, Alejandro Dominguez Rodriguez, Full time professor of Psychology, Universidad Autonoma de Baja California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F-PROMEP-38/Rev-04
Record Dates: First submitted 2019-04-08; First posted 2019-04-16 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Anxiety Disorders
Keywords: General Anxiety Disorder; Social Anxiety Disorder; Specific Phobia; Obsessive Compulsive Disorder; posttraumatic stress disorder
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder; Phobia, Social; Phobia, Specific; Obsessive-Compulsive Disorder; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: The study has two arms, one is the intervention group that receive the treatment and the other is the control group that does not receive treatment, just waiting list, however at the end of the assesment the participants in the control group will also receive the treatment. The patients in both groups will be evaluated pre and post treatment. 11 sessions, once per week, therefore 3 months apart.
Who Masked: Participant
Masking Description: The patients are not aware that there is an intervention group and a control group, the participants are not related and do not know each other. The conditions of the study are only known by the researcher, the therapists and the bioethics committee of the Autonomous University of Baja California. The participants are assigned randomly to the intervention or control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transdiagnostic Treatment (Experimental): Participants in this group will receive from 11 to 17 sessions of the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders.
  Interventions: Behavioral: Transdiagnostic Treatment
- Control group (No Intervention): The participants in this group will not receive the treatment, just waiting list. They will be measured one time and then a second time 3 months after. Calculating when 3 months corresponding to 11-12 sessions will take place in the intervention group.

INTERVENTIONS:
Behavioral: Transdiagnostic Treatment — The Unified Transdiagnostic Protocol (PUT) is a cognitive-behavioral treatment focused on emotions. "The PUT was developed to be applicable to anxiety disorders, mood disorders, as well as other disorders in which anxiety and emotional dysregulation play an important role, such as many somatoform and dissociative disorders".
  The PUT proposal includes 8 modules, of which 5 are nuclear, it is recommended to give these modules between 11 to 17 sessions with a duration of one hour each.
  Arms: Transdiagnostic Treatment

SUMMARY:
This study evaluates the effectiveness of The Unified Transdiagnostic Protocol, a psychological treatment for the intervention of a broad range of anxiety disorders. It is compared the effectiveness of the treatment with the changes of the same participants before and after the treatment and a control group. The changes are being assessed through subjective measures such as psychometrics and objective measures such as Electroencelophalography.

DETAILED DESCRIPTION:
Anxiety disorders are among the highest prevalence of disorders in the general population worldwide, however, in the last decades they were treated by separate.

However, it has been proposed that several emotional disorders have a common root and can be treated similarly. This is called the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders. The treatment has as objective to be implemented from 11 to 17 sessions, with 8 modules. This treatment can be applied to a bigger range of disorders, not only anxiety disorder, however, the objective of this study is to focus on the most urgent disorders in the border of Mexico and USA, that are anxiety disorders. According to the available scientific literature, this is the first time that this study has been applied in Mexican population. This study will have an intervention group that will receive the transdiagnostic treatment, and a control group that will be in a waiting list, and after the waiting list and the measured took place these patients will also receive the treatment. In both conditions the participants will be measured pre and post. The subjective measures will include the following psychometrics:

1. Post-Traumatic Stress Disorder (PTSD) Symptom Scale (PSS).
2. Interview Program for Anxiety Disorders.
3. Beck Depression Inventory.
4. State Trait Anxiety Inventory.
5. Generalized Anxiety Disorder 7-item (GAD-7) scale .
6. Big Five Inventory.
7. Scale of Beck's Suicidal Ideation.
8. Yale-BrownObsessive Compulsive Scale (Y-BOCS)

Also it is planned to measure the brain activity through an electroencephalogram, specifically the Gamma rhythm. It has been observed that when patients with General Anxiety disorder are emotionally aroused their Gamma rhythm increases. Part of the objectives of this study is to replicate the procedure by Oathes et al., that consist in measuring the brain activity of the participants with an electroencephalogram of 17 channels, following these steps: 2 minutes' base line, 5 minute relaxation and 5 minutes emotionally aroused, in their study it was observed in the patients that the Gamma rhythm was lower in the relaxation phase, increasing at the base line and having the highest record in the emotionally aroused minutes. To perform this measure, it will be used the EMOTIVE EPOC + of 14 channels is non-invasive, painless, low cost method Used for scientific research. The 14 channels with which the device counts. It allows to measure the cerebral areas AF3, F7, F3, FC5, T7, P7, O1, O2, P8, T8, FC6, F4, F8, AF4, based on the international system 10-20.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of General Anxiety Disorder and/or Panic Disorder and/or Posttraumatic Stress Disorder and/or Social Anxiety Disorder and / or Obsessive Compulsive Disorder.

Exclusion Criteria:

* Consuming drugs
* To receive another psychological treatment in the same period of the study
* To be consuming medicines to treat symptoms of anxiety or depression
* To show comorbidity with a psychiatric disorder
* Moderate to high score in the suicide scale
* Recent attempt of suicide (3 months) measured with the Scale of Beck's Suicidal Ideation (Beck, Steer and Ranieri, 1988).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Decrease in the scores of the Post-Traumatic Stress Disorder Symptom Scale | 3 to 4.5 months, depending on the development of the patient and the sessions needed, 11 to 17.
  The Post-Traumatic Stress Disorder Symptom Scale is a 17-item structured interview. The severity over the last 2 weeks of each item on the PSS is rated by the interviewer using a 4-point scale: 0 = not at all, 1 = a little bit, 2 = somewhat, and 3 = very much. The maximum possible score is 51 (severely affected) and the minimum possible score is 0 (total absence of the symptoms). The total severity score is calculated as the sum of the severity ratings for the 17 items. The diagnosis of the Post-Traumatic Stress Disorder Symptom Scale is made when at least 1 re-experiencing, 3 avoidance and 2 arousal symptoms are endorsed on the scale by individuals who were traumatized at least one month prior to the assessment. It is expected a statistical significant decrease (P < 0.05) in the symptoms of Post-Traumatic Stress Disorder in the patients suffering from this disorder.
Decrease in the score of Anxiety symptoms | 3 to 4.5 months, depending on the development of the patient and the sessions needed, 11 to 17.
  The State Trait Anxiety Inventory consists of two subscales of 20 items each that measure anxiety as a transient state of tension (Scale A-State), and as a characteristic of the personality relatively stable over time (Scale B -trait). The items are composed by an assertion to which the subject responds indicating their degree of identification. In the case of state anxiety, the scale goes from 1 (not at all), 2 (somewhat), 3 (moderately), 4 (very much), while in the trait anxiety it ranges from 1 (almost never), 2 (sometimes), 3 (often), 4 (almost always). In both, a percentage of the items evaluates well-being or absence of anxiety, while the rest of the items to the presence of anxiety. Scores range from 20 to 80, in each subscale, with higher scores correlating with greater anxiety. It is expected a statistical significant decrease (P < 0.05) in the anxiety symptoms.
Decrease in the symptoms of depression | 3 to 4.5 months, depending on the development of the patient and the sessions needed, 11 to 17.
  The Beck Depression Inventory is a self-report that provides a measure of the presence and severity of depression. Contains 21 items indicative of symptoms such as sadness, crying, loss of pleasure, feelings of failure and guilt, suicidal thoughts or desires, pessimism, etc. Each item is answered on a 4-point scale, from 0 to 3, where each number is identified different for each item, in all of them 0 means absence and 3 full presence (e.g. sadness), except for items 16 (changes in the sleep pattern) and 18 (changes in appetite) that contain 7 categories. The minimum and maximum scores in the test are 0 and 63. Cut-off points ha that allow to classify those evaluated in one of the following four groups: 0-13, minimum depression; 14-19, mild depression; 20-28, moderate depression; and 29-63, severe depression. It is expected a statistical significant decrease (P < 0.05) in the depression symptoms.
Decrease in the symptoms of General Anxiety Disorder | 3 to 4.5 months, depending on the development of the patient and the sessions needed, 11 to 17.
  On the Generalized Anxiety Disorder 7-item (GAD-7) scale subjects are asked how often, during the last 2 weeks, they have been bothered by each of the 7 core symptoms of generalized anxiety disorder. Response options are "not at all," "several days," "more than half the days," and "nearly every day," scored as 0, 1, 2, and 3, respectively. Therefore, GAD-7 scores range from 0 to 21, with scores of ≥5, ≥10, and ≥15 representing mild, moderate, and severe anxiety symptom levels, respectively. It is expected a statistical significant decrease (P < 0.05) in the General Anxiety symptoms.
Decrease in gamma rhythm measures | 3 to 4.5 months, depending on the development of the patient and the sessions needed, 11 to 17.
  Decrease in the gamma rhythm trough the EEG measure. The decrease will be shown comparing the participants in the intervention group within their own results in the pre to post measures, and comparing the participants in the control group vs. the intervention group.
Decrease is Obsessive Compulsive symptoms | 3 to 4.5 months, depending on the development of the patient and the sessions needed, 11 to 17.
  The Yale-BrownObsessive Compulsive Scale (Y-BOCS) is composed of 10 items: 5 related to obsessions and the other 5, to compulsions, having an answer option from 0 to 4 (from not presenting a symptom until presenting extreme symptoms). The diagnostic classification is based on the points of cut where 0 to 7 represents "without clinical manifestations", 8 to 15, "mild", 16 to 23, "moderate", 24 to 31 as "severe" and 32 to 40 as "extreme". It is expected a statistical significant decrease (P < 0.05) in the Obsesive Compulsive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Dominguez-Rodriguez, PhD, Study Director — Autonomous University of Baja California
Locations (2):
- Mexico (2):
  - Universidad Autonoma de Ciudad Juarez, Juárez, Chihuahua
  - Autonomous University of Baja California, Tijuana, Estado de Baja California

IPD SHARING:
Plan to Share IPD: Yes
The information will be available in a private server or in a server of the journal(s) that we will publish the articles that will be the result of this study. The protocol of the study is currently in progress to be published, in this article will be included such study protocol, statistical analysis plan and the informed consent is already shared in the register of clinical trials.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: This data will be available approximately in January 2020 and it will be permanently available. It wil be shared in the databases of the journal where the article(s) will be published
Access Criteria: Through the servers of the journal(s) where we will publish the articles.

REFERENCES:
- [Background] Beck AT, Steer, RA, Brown, GK. Manual for Beck Depression Inventory-II. (1996) San Antonio, TX: Psychological Corporation.
- [Background] Beck AT, Steer RA, Ranieri WF. Scale for Suicide Ideation: psychometric properties of a self-report version. J Clin Psychol. 1988 Jul;44(4):499-505. doi: 10.1002/1097-4679(198807)44:43.0.co;2-6. PMID 3170753
- [Background] Brown TA, Di Nardo PA, Lehman CL, Campbell LA. Reliability of DSM-IV anxiety and mood disorders: implications for the classification of emotional disorders. J Abnorm Psychol. 2001 Feb;110(1):49-58. doi: 10.1037//0021-843x.110.1.49. PMID 11261399
- [Background] Ellard KK, Fairholme CP, Boisseau CL, Farchione TJ, Barlow DH. Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders: Protocol Development and Initial Outcome Data. Cogn Behav Pract. 2010 Feb;17(1):88-101. doi: 10.1016/j.cbpra.2009.06.002. Epub 2010 Jan 29. PMID 33762811
- [Background] Foa EB, Cashman L, Jaycox L, Perry K. The validation of a self-report measure of posttraumatic stress disorder: The posttraumatic diagnostic scale. Psychol Assess 1997;9(4):445-451.
- [Background] Goodman WK, Price LH, Rasmussen SA, Mazure C, Fleischmann RL, Hill CL, Heninger GR, Charney DS. The Yale-Brown Obsessive Compulsive Scale. I. Development, use, and reliability. Arch Gen Psychiatry. 1989 Nov;46(11):1006-11. doi: 10.1001/archpsyc.1989.01810110048007. PMID 2684084
- [Background] John OP, Naumann LP, Soto CJ. Paradigm Shift to the Integrative Big-Five Trait Taxonomy: History, Measurement, and Conceptual Issues. In O. P. John, R. W. Robins, & L. A. Pervin (Eds.), Handbook of personality: Theory and research (pp. 114-158). 2008 New York, NY: Guilford Press.
- [Background] Kennedy KA, Barlow DH. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders: An introduction. In Farchione TJ, Barlow, DH (Eds.), Applications of the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders. New York: Oxford University Press. 2017
- [Background] Oathes DJ, Ray WJ, Yamasaki AS, Borkovec TD, Castonguay LG, Newman MG, Nitschke J. Worry, generalized anxiety disorder, and emotion: evidence from the EEG gamma band. Biol Psychol. 2008 Oct;79(2):165-70. doi: 10.1016/j.biopsycho.2008.04.005. Epub 2008 Apr 15. PMID 18499328
- [Background] Spielberger C, Diaz-Guerrero R. IDARE: Inventario de Ansiedad Rasgo-Estado. México: Manual Moderno. 1975
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Yacila GA, Cook-del Aguila L, Sanchez-Castro AE, Reyes-Bossio M, Tejada RA. Traducción y adaptación cultural del Yale-Brown Obsessive Compulsive Scale (Y-BOCS) para trastornos obsesivos compulsivos Spanish translation and cultural adaptation of Yale- Brown Obsessive Compulsive Scale (Y-BOCS). Acta Médica Peruana. 2016. 33 (3):253-255.
- [Background] Lowe B, Decker O, Muller S, Brahler E, Schellberg D, Herzog W, Herzberg PY. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. Med Care. 2008 Mar;46(3):266-74. doi: 10.1097/MLR.0b013e318160d093. PMID 18388841
- [Background] Hishinuma ES, Miyamoto RH, Nishimura ST, Nahulu LB, Andrade NN, Makini GK Jr, Yuen NY, Johnson RC, Kim SP, Goebert DA, Guerrero AP. Psychometric properties of the state-trait anxiety inventory for Asian/Pacific-islander adolescents. Assessment. 2000 Mar;7(1):17-36. doi: 10.1177/107319110000700102. PMID 10668003
- See also: EMOTIV Epoc + 14 Channel Wireless EEG Headset. (2019, April). — https://www.emotiv.com/epoc/

DOCUMENTS (1):
  • Informed Consent Form (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT03916315/ICF_000.pdf